CLINICAL TRIAL: NCT00881569
Title: Extended Use of CS 7017 Upon Completion of Participation in a Clinical Study of CS-7017 in Subjects With Cancer
Brief Title: Extended Use Protocol for Participants With Cancer to Receive Continued Treatment With CS-7017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-U102E
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Advanced Cancer
Keywords: CS-7017; Advanced Cancer
MeSH Terms: interventions — efatutazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CS-7017 tablets twice daily at strength ranging from 0.5 mg to 0.75 mg
  Interventions: Drug: CS-7017

INTERVENTIONS:
Drug: CS-7017 — CS-7017 administered orally, twice daily continuously for 6 weeks

SUMMARY:
This is a study of CS-7017 designed to allow participants who completed participation in a clinical study of CS-7017 without experiencing disease progression or unacceptable toxicity to continue treatment with study drug. Participants who have not progressed while receiving CS-7017 will continue to benefit from longer administration of the agent.

DETAILED DESCRIPTION:
This is an open-label non-randomized study of CS-7017 designed to allow participants who completed participation in a clinical study of CS-7017 without experiencing disease progression or unacceptable toxicity to continue treatment with study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant previously treated with CS-7017 as part of a study that included CS-7017 and has shown clinical benefits from treatment with CS-7017.

Exclusion Criteria:

* Anticipation of need for a major surgical procedure or radiation therapy during the study.
* Any of the following conditions within 6 months prior to initiating study treatment: Myocardial infarction with significant impairment of cardiac function (eg, ejection fraction ≤ 50%), severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class II or higher congestive heart failure.
* Participants with clinically significant pleural or pericardial effusions.
* Clinically significant active infection, which requires antibiotic therapy, or human immune deficiency virus (HIV)-positive subjects receiving antiretroviral therapy.
* Participants with diabetes mellitus requiring treatment with insulin, sulfonylureas or thiazolidinediones (TZDs) agents, malabsorption syndrome, chronic diarrhea, inflammatory bowel disease, or partial bowel obstruction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2 participants who met all inclusion and no exclusion criteria were enrolled in this extension study at 1 clinic site in the United States.
Pre-assignment Details: This extension study was designed to allow continuation of treatment in participants who demonstrated clinical benefit from previous treatment with CS-7017 in CS7017-A-U102 study.
Groups:
- CS-7017 0.75 mg BID: Participant who received oral CS-7017 0.75 mg twice daily (BID).
- CS-7017 0.50 mg BID: Participant who received oral CS-7017 0.50 mg twice daily (BID).
Period: Overall Study
Arm/Group | CS-7017 0.75 mg BID | CS-7017 0.50 mg BID
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Disease progression | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-7017 0.50 mg BID | CS-7017 0.75 mg BID | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (0) | 42 (0) | 57 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Best Response Following Extended Use of CS-7017 Upon Completion of Participation in a Clinical Study of CS-7017 in Participants With Cancer
Description: At each evaluation, the participant's status was assessed as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD); the best response was then identified. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions).
Time Frame: From baseline and every 6 weeks postdose, up to 2 years 6 months
Population: Best response was assessed in All Enrolled Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.50 mg BID | CS-7017 0.75 mg BID
Number analyzed (Participants) | 1 | 1
Participants
  Partial response (PR) | 0 | 1
  Stable disease (SD) | 1 | 0

2. Secondary Outcome: Response/Stable Disease Duration and Time to Progression Following Extended Use of CS-7017 Upon Completion of Participation in a Clinical Study of CS-7017 in Participants With Cancer
Description: Duration of response was to be calculated as the date of progression minus the earliest date of complete response (CR) or partial response (PR), plus 1. The earliest date of CR or PR was to be taken from the earlier study (CS7017-A-U102). If any participant entered the study with stable disease (SD), then the duration of SD was to be calculated as the date of progression minus the date of first dose, plus 1. Time to progression was to be calculated as the date of progression minus the date of first dose of study medication in the earlier study, plus 1.
Time Frame: Baseline and every 6 weeks postdose, up to 2 years 6 months
Population: Duration of response/stable disease and time to progression were assessed in All Enrolled Participants.
Measure: Number; unit: days
Arm/Group | CS-7017 0.50 mg BID | CS-7017 0.75 mg BID
Number analyzed (Participants) | 1 | 1
days
  Response duration | NA — A complete response or partial response was not observed in this participant; therefore, this assessment was not applicable. | 441
  Time to progression | 337 | 686
  Stable disease duration | 337 | NA — Stable disease was not observed in this participant; therefore, this assessment was not applicable.

3. Secondary Outcome: Treatment-Emergent Adverse Events Occurring in Participants Following Extended Use of CS-7017 Upon Completion of Participation in a Clinical Study of CS-7017 in Participants With Cancer
Description: Adverse events (AEs) were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0. AE intensity was assessed according to the following scale: Mild (Grade 1), Awareness of sign or symptom, but easily tolerated, ie, does not interfere with subject's usual function; Moderate (Grade 2), Discomfort enough to cause interference with usual activity; Severe (Grade 3), Incapacitating with inability to work or do usual activity, ie, interferes significantly with participant's usual function. Severe (Grade 3) AEs indicate worse outcomes.
Time Frame: Baseline up to 30 days after last dose, up to 2 years 6 months
Population: Safety events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.50 mg BID | CS-7017 0.75 mg BID
Number analyzed (Participants) | 1 | 1
Participants
  Grade 3 Hypercholesterolemia | 0 | 1
  Grade 1-2 Hypertriglyceridemia | 0 | 1
  Grade 1 Fatigue | 0 | 1
  Grade 3 Anaemia | 1 | 0
  Grade 1-2 Anaemia | 1 | 0
  Grade 1 Regurgitation | 1 | 0
  Grade 1 Tongue paralysis | 1 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days after last dose, up to 2 years 6 months.
Description: A treatment-emergent adverse event (TEAEs) was defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the first dose until 30 days after the last dose.
Arm/Group | CS-7017 0.50 mg BID | CS-7017 0.75 mg BID
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.50 mg BID (N=1) | CS-7017 0.75 mg BID (N=1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglceridemia (Metabolism and nutrition disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Tongue paralysis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No